CLINICAL TRIAL: NCT01101971
Title: Can a MEdTech E-learning Module Adequately Prepare Medical Students to Undertake a First Female Pelvic Exam?
Brief Title: Preparing Medical Students to Undertake a First Female Pelvic Exam.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Robert Reid, Principal Investigator, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OBGY-199-10
Record Dates: First submitted 2010-04-08; First posted 2010-04-12 (Estimated); Results first posted 2017-06-16 (Actual); Last update posted 2017-06-16 (Actual); Status verified 2017-04

CONDITIONS: Female Pelvic Exam
Keywords: Education, Medical; Students, Medical; Gynecology; Physical Examination; Computer-Assisted Instruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- first year medical students (Experimental)
  Interventions: Other: Pelvic exam video tutorial

INTERVENTIONS:
Other: Pelvic exam video tutorial — Bryden Magee (Meds 2010) and Dr. Robert Reid created an educational DVD © 2009 that outlines a step-by-step approach to the pelvic exam; utilizing real patient video clips and illustrations. Endorsed by the Association of Professors of Obstetrics and Gynaecology of Canada (APOG), this innovation has been shown to improve both knowledge and confidence in medical students learning these skills (Magee 2009). The video content has been posted on the Queen's streaming server and incorporated into a MEdTech community accessible to all Queen's faculty and students affiliated with the School of Medicine (in MEdTech Central see OBGYN Pelvic Exam Module under community courses).
  Other Names: Educational DVD © 2009

SUMMARY:
Objective: To evaluate the effectiveness of a web based learning module in the preparation of medical students to undertake a first female pelvic exam.

Background: Bryden Magee (Meds 2010) under the supervision of Robert Reid, M.D., created an educational DVD © 2009 that gives a step-by-step approach to the pelvic exam utilizing real patient video clips and illustrations. Endorsed by the Association of Professors of Obstetrics and Gynaecology of Canada (APOG), this educational innovation has been shown to improve both knowledge and confidence in medical students learning these skills (Magee 2009). The video content is accessible to all Queen's faculty and students affiliated with the School of Medicine through MEdTech.

Methods: We will introduce medical students to the MEdTech pelvic exam module and use a comprehensive assessment tool, designed by experienced gynaecologists in our Department, to measure how well they perform their first exam on female volunteers acting as mock patients. We plan to recruit 48 students and 4 mock patients.

Outcome: We will evaluate the success rate of students achieving a passing grade of 50% (12/24) on their first unassisted speculum and bimanual examination after viewing the video content.

DETAILED DESCRIPTION:
At Queen's University students may have many months between their gynaecology teaching associates (GTAs) teaching session and their first attendance at gynaecology clinics. In many circumstances their preparedness to perform a first examination seems limited. The first examination experience in clinic is the most critical since subsequent examinations are done after critique and feedback. We wish to determine whether our web-based video instruction module, when viewed immediately prior to the first examination, adequately prepares naïve students to skilfully perform their first pelvic exam. This will require simulated patients, qualified examiners, and the use of a comprehensive assessment tool. If this technology is effective this will offer significant savings in terms of time to the medical school for scheduling of many GTAs sessions over many months, to the students who currently set aside two hours for a GTA session, and in terms of ongoing costs ($200 per student for GTA sessions; $20,000 per year).

Objective: To evaluate the effectiveness of a MEdTech e-learning module designed to prepare medical students to undertake a first female pelvic exam.

Methods: We will introduce first year medical students to the MEdTech e-learning module. Following this exposure we will measure how well they perform their first exam on female volunteers acting as mock patients using a comprehensive 23-item assessment tool designed by experienced gynaecologists in our Department.

We will recruit four women to act as simulated patients. We are expecting that 48 students will choose to participate in our study. Four residents from the Department of Obstetrics and Gynaecology will act as examiners. We estimate it will take 20 minutes for each student to perform a pelvic exam, and to be graded and receive feedback by a resident examiner. Four exams per simulated patient would allow our research team to test 48 students over three sessions. The study will take place in the Fraser Armstrong Patient Centre of the Kingston General Hospital which has the requisite examination rooms and examination equipment. The nursing supervisor (Donna Cooper) has given approval to this educational research protocol.

To troubleshoot logistics we will run a small pilot study with four students and four simulated patients. This session will also serve to provide instructions to the mock patients and to validate our scoring system.

Limitations: Our design does not incorporate a comparison group, which would logically be third year medical students exposed to the current curriculum which incorporates GTAs. The aim of such a noninferiority trial would be to show that our web-based educational module is not inferior to the current teaching standard. Anticipating an overall pass rate of 80% and using a margin of indifference of 10%, 253 students would be required per group; 80% Power; 5% alpha level (Pocock 2003). Recognizing that this sample size is clearly not feasible; we have elected to go with this non-comparative design. We believe this study will provide relevant data that can be applied to our medical education curricula, possibly resulting in substantial savings of both time and cost.

ELIGIBILITY:
Inclusion Criteria:

* Year one of medical school

Exclusion Criteria:

* Any previous clinical training in performing pelvic exams

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2010-04; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert L Reid, M.D., Principal Investigator — Queen's University
Locations (1):
- Fraser Armstrong Patient Clinic, Kingston General Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Beckmann CR, Lipscomb GH, Williford L, Bryant E, Ling FW. Gynaecological teaching associates in the 1990s. Med Educ. 1992 Mar;26(2):105-9. doi: 10.1111/j.1365-2923.1992.tb00134.x. PMID 1565025
- [Background] Magee B, Hahn P, Reid RL. The comprehensive female pelvic examination educational DVD: Improving knowledge and confidence in medical students. [Abstract] J Obstet Gynaecol Can 2009 Jan;31(1):74-5.
- [Background] Orientale E Jr, Kosowicz L, Alerte A, Pfeiffer C, Harrington K, Palley J, Brown S, Sapieha-Yanchak T. Using web-based video to enhance physical examination skills in medical students. Fam Med. 2008 Jul-Aug;40(7):471-6. PMID 18928073
- [Background] Pickard S, Baraitser P, Rymer J, Piper J. Can gynaecology teaching associates provide high quality effective training for medical students in the United Kingdom? Comparative study. BMJ. 2003 Dec 13;327(7428):1389-92. doi: 10.1136/bmj.327.7428.1389. PMID 14670887
- [Background] Pocock SJ. The pros and cons of noninferiority trials. Fundam Clin Pharmacol. 2003 Aug;17(4):483-90. doi: 10.1046/j.1472-8206.2003.00162.x. PMID 12914552

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First-year medical students, excluding any with previous clinical training in performing pelvic examinations, were recruited to participate in this study.
Period: Overall Study
Arm/Group | First Year Medical Students
Started | 45
Completed | 45
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | First Year Medical Students
Number analyzed (Participants) | 45
Age, Continuous [Mean (Full Range); unit: years] | 24 [20 to 40]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 23
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 45

OUTCOME MEASURES:

1. Primary Outcome: Score on Pelvic Exam Assessment Tool
Description: A pelvic exam assessment score out of 30 is recorded by a Resident examiner immediately after a student completes their first pelvic examination on a mock patient. Pass = 15/30 (50%).
Time Frame: 15 minutes
Measure: Mean (Standard Deviation); unit: points
Arm/Group | First Year Medical Students
Number analyzed (Participants) | 45
points | 23.9 (3.9)

ADVERSE EVENTS:
Arm/Group | First Year Medical Students
All-Cause Mortality (participants affected / at risk) | 0/45
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 0/45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes